CLINICAL TRIAL: NCT01148303
Title: Randomized, Placebo Controlled Trial of Etoricoxib (Arcoxia) Taken Prophylactically to Prevent Ramadan Headache
Brief Title: Trial of Etoricoxib (Arcoxia) Taken Prophylactically to Prevent Ramadan Headache
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hartford Hospital (Other)
Collaborators: Shaare Zedek Medical Center (Other)
Responsible Party: Michael J Drescher MD, Hartford Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: ARX_ISP_IL1001
Record Dates: First submitted 2010-06-17; First posted 2010-06-22 (Estimated); Last update posted 2011-03-08 (Estimated); Status verified 2011-03

CONDITIONS: Headache; Fasting; Fasting Headache; Ramadan Headache
Keywords: Headache; Fasting; Fasting Headache; Ramadan; Ramadan Headache; Yom Kippur; Yom Kippur Headache
MeSH Terms: conditions — Headache; Fasting | interventions — Etoricoxib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Etoricoxib First (Experimental): This arm will receive etoricoxib for six days, followed by placebo for eight days.
  Interventions: Drug: Etoricoxib; Drug: Placebo
- Etoricoxib Second (Experimental): This arm will get placebo for eight days before beginning their fast, followed by etoricoxib for six days.
  Interventions: Drug: Etoricoxib; Drug: Placebo

INTERVENTIONS:
Drug: Etoricoxib — Subjects will take etoricoxib 90mg by mouth just before the start of the daily fast. This will be for six days. After this they will receive placebo for eight days.
  Other Names: arcoxia
  Arms: Etoricoxib First
Drug: Etoricoxib — This arm will receive placebo just before their fast for eight days. After this they will receive etoricoxib 90mg just before their daily fast for the next six days.
  Other Names: Arcoxia
  Arms: Etoricoxib Second
Drug: Placebo — Placebo

SUMMARY:
The investigators intend to study whether the use of the pain medication etoricoxib (Arcoxia) taken just before the Ramadan fast will prevent or lessen headache that some people get while fasting. The investigators hypothesize that etoricoxib will reduce the number of people getting headache, more than placebo. The investigators will do this by giving participants in the study either real medication or placebo (sugar pill) and comparing the results. The investigators will study this over two weeks. The first week one group will get the medicine and the other the placebo. The second the groups will switch. Neither the subjects nor the investigators will know who is in which group.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 -65.
* Patients will be enrolled if they declared that they intended to complete the dawn to dusk Ramadan fast, and had demonstrated their commitment by doing so for the previous three years (unless medically prevented.)
* Patient states that he/she typically suffered from headache during fasting in the past.

Exclusion Criteria:

* Patients with a history of severe cardiovascular disease, diabetes, asthma, COPD, hypertension, or a history of bleeding, particularly in the gastrointestinal tract
* Patients who have experienced bronchospasm, acute rhinitis, nasal polyps, angioneurotic oedema, urticaria, or allergic-type reactions after taking acetylsalicylic acid or NSAIDs including COX-2 (cyclooxygenase-2) inhibitors
* Pregnant or lactating patients. Sexually active women of childbearing age will be included only if using birth control
* Severe hepatic dysfunction
* Estimated renal creatinine clearance <30 ml/min
* History of peptic ulcer, erosive gastritis, esophagitis or inflammatory bowel disease
* Congestive heart failure
* Patients with hypertension whose blood pressure is persistently elevated above 140/90mmHg and has not been adequately controlled Established ischaemic heart disease, peripheral arterial disease, and/or cerebrovascular disease
* Cancer or any other malignant disease
* History of medication overuse. Overuse of analgesics or antimigraine drugs according to the IHS criteria (chapter 8)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2010-07; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Headache | Two weeks
  The subjects will be asked to fill out a daily 'headache diary' at the end of the fast. They will be asked if they had a headache on that day, and if so its severity. We will then compare the number of subjects having a headache on each day and total number of 'headache days' between the groups.

SECONDARY OUTCOMES:
Severity of Headache | Two weeks
  We will ask the subject if they had a headache on a given day to rate its severity. We will then compare the severity of headache between groups.
Overall ease of fast | Two weeks
  We will ask subjects to rate the ease of their fast on a daily basis on a 5 point scale and will compare general ease of fast between the groups.
Side effects and other symptoms | two weeks
  We will ask subjects to record other symptoms or side effects they had during the fast including nausea, abdominal pain, photophobia, difficulty breathing or other.

CONTACTS AND LOCATIONS:
Overall Officials: Naim Shehadeh, MD, Principal Investigator — Rambam Health Care Campus; Zev Wimpfheimer, MD, Principal Investigator — Shaare Zedek Medical Center
Locations (1):
- Shaare Zedek Medical Center, Jerusalem, Israel

REFERENCES:
- [Background] Drescher MJ, Elstein Y. Prophylactic COX 2 inhibitor: an end to the Yom Kippur headache. Headache. 2006 Nov-Dec;46(10):1487-91. doi: 10.1111/j.1526-4610.2006.00609.x. PMID 17115981
- [Background] Drescher MJ, Alpert EA, Zalut T, Torgovicky R, Wimpfheimer Z. Prophylactic etoricoxib is effective in preventing Yom Kippur headache: a placebo-controlled double-blind and randomized trial of prophylaxis for ritual fasting headache. Headache. 2010 Sep;50(8):1328-34. doi: 10.1111/j.1526-4610.2009.01587.x. Epub 2009 Dec 21. PMID 20039959
- [Background] Topacoglu H, Karcioglu O, Yuruktumen A, Kiran S, Cimrin AH, Ozucelik DN, Sarikaya S, Soysal S, Turpcu U, Bozkurt S. Impact of Ramadan on demographics and frequencies of disease-related visits in the emergency department. Int J Clin Pract. 2005 Aug;59(8):900-5. doi: 10.1111/j.1742-1241.2005.00460.x. PMID 16033610
- [Background] Awada A, al Jumah M. The first-of-Ramadan headache. Headache. 1999 Jul-Aug;39(7):490-3. doi: 10.1046/j.1526-4610.1999.3907490.x. PMID 11279933
- [Background] Shah PA, Nafee A. Clinical profile of headache and cranial neuralgias. J Assoc Physicians India. 1999 Nov;47(11):1072-5. PMID 10862316
- [Derived] Drescher MJ, Wimpfheimer Z, Abu Khalef S, Gammaitoni A, Shehadeh N, Torgovicky R. Prophylactic etoricoxib is effective in preventing "first of Ramadan" headache: a placebo-controlled double-blind and randomized trial of prophylactic etoricoxib for ritual fasting headache. Headache. 2012 Apr;52(4):573-81. doi: 10.1111/j.1526-4610.2011.01993.x. Epub 2011 Aug 16. PMID 21848948